CLINICAL TRIAL: NCT05118282
Title: A Coping Skills Program for Children With Asthma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017-04-0128
Record Dates: First submitted 2021-10-14; First posted 2021-11-11 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Asthma in Children

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combined coping skills + asthma management arm (Experimental): The combined coping skills + asthma management arm is a family-based coping skills + asthma management intervention that is bilingual and culturally relevant for Latino families. This program is manualized with video-guided and interactive content to improve coping with stress and asthma management behaviors for both children and their parents. Coping strategies taught include primary and secondary control coping. Asthma management content is interactive and culturally tailored.
  Interventions: Behavioral: Combined coping skills + asthma management
- Standard asthma management arm (Active Comparator): The standard asthma management (AM) arm is an asthma management intervention covering standard asthma self-management content (e.g., symptom recognition, self-monitoring). AM is manualized and is matched in length, time, and number of sessions to the experimental arm.
  Interventions: Behavioral: Standard Asthma Management (AM)

INTERVENTIONS:
Behavioral: Combined coping skills + asthma management — This arm includes a curriculum teaching coping skills and culturally relevant asthma management skills.
  Arms: Combined coping skills + asthma management arm
Behavioral: Standard Asthma Management (AM) — This arm includes a curriculum teaching standard asthma management skills.
  Arms: Standard asthma management arm

SUMMARY:
Uncontrolled asthma in school-aged children is a significant public health problem. Latino children living in low-income contexts are at increased risk for uncontrolled asthma compared to non-Latino white children, and stress is an unaddressed factor in this disparity. Therefore, the purpose of the current study is to test an intervention program that teaches families skills to cope with asthma-related and other sources of stress. Specifically, the study will compare the effects of the combined coping skills + asthma management program with a standard asthma management program in 280 families of Latino children with asthma. The study will also look at why the program may have an effect, and specifically whether the program impacts child coping, parent coping, or family asthma management behaviors. The main hypothesis is that the combined coping skills + asthma management program will improve asthma outcomes more than the standard asthma management program.

DETAILED DESCRIPTION:
This study is a randomized controlled trial (RCT) examining the effects and mediators of Adapt 2 Asthma (A2A), a coping skills + asthma management intervention, compared to standard asthma self-management (AM) for Latino children with asthma and their parents/caregivers living in low-socioeconomic status (SES) contexts. The focus of the study is to test the effects of A2A on asthma control, quality of life, lung function, school absences, and emergency department visits, and to identify child and parent mediational pathways of A2A.

Children ages 8 to 14 years old with asthma and their parents/caregivers will participate. The investigators will enroll 280 youth who are patients at the partner primary care clinics and 280 of their parents/caregivers to participate. The investigators will identify patients with asthma in the study age range through reviewing records from the partner clinics as well as natural referral when patients attend appointments. The investigators will screen identified patients for eligibility. Enrolled families will complete assessments at 1 week pre-intervention, 1 week post-intervention, and at 6- and 12-month follow-up timepoints.

Research staff will collect assessment data in the form of child and parent surveys, interviews and spirometry. Providers will also audiotape sessions, which will be used for case supervision and to measure fidelity to the intervention. Youth and parents/caregivers will provide all data. Participant data will be de-identified and stored in the principal investigator's locked laboratory, and all computerized data will be encrypted with University approved encryption software to ensure the confidentiality, integrity and availability of data.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria are that (a) the child has a diagnosis of asthma as reported by the child's medical provider and confirmed by the parent; (b) the child is a current patient at a participating clinic; (c) the child is 8 to 14 years old; (d) the child is Latino/a; and (e) the child and parent speak English or Spanish.

Exclusion Criteria:

* Exclusion criteria are that the presence of a disability interferes with the child's participation in the intervention beyond accommodations feasible in primary care.

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 560 (Estimated)
Dates: Start 2021-11-14 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Asthma Control as measured by the Asthma Control Test (ACT) | Baseline
  The Asthma Control Test assesses symptom control and impairment due to asthma (e.g., "how often have you had shortness of breath"). The ACT has versions for children ages 4-11 and 12 and older and is responsive to clinical change.
Asthma Control as measured by the Asthma Therapy Assessment Questionnaire (ATAQ) | Baseline
  The Asthma Therapy Assessment Questionnaire (cATAQ) is a parent-report questionnaire; the symptom control subscale assesses children's asthma control (e.g., "wheezing or difficulty breathing") and shows good reliability and validity.
Asthma Control as measured by the Asthma Control Test (ACT) | 1 week Post-intervention
  The Asthma Control Test assesses symptom control and impairment due to asthma (e.g., "how often have you had shortness of breath"). The ACT has versions for children ages 4-11 and 12 and older and is responsive to clinical change.
Asthma Control as measured by the Asthma Therapy Assessment Questionnaire (ATAQ) | 1 week Post-intervention
  The Asthma Therapy Assessment Questionnaire (cATAQ) is a parent-report questionnaire; the symptom control subscale assesses children's asthma control (e.g., "wheezing or difficulty breathing") and shows good reliability and validity.
Asthma Control as measured by the Asthma Control Test (ACT) | 6 months post-intervention
  The Asthma Control Test assesses symptom control and impairment due to asthma (e.g., "how often have you had shortness of breath"). The ACT has versions for children ages 4-11 and 12 and older and is responsive to clinical change.
Asthma Control as measured by the Asthma Therapy Assessment Questionnaire (ATAQ) | 6 months post-intervention
  The Asthma Therapy Assessment Questionnaire (cATAQ) is a parent-report questionnaire; the symptom control subscale assesses children's asthma control (e.g., "wheezing or difficulty breathing") and shows good reliability and validity.
Asthma Control as measured by the Asthma Control Test (ACT) | 12 months post-intervention
  The Asthma Control Test assesses symptom control and impairment due to asthma (e.g., "how often have you had shortness of breath"). The ACT has versions for children ages 4-11 and 12 and older and is responsive to clinical change.
Asthma Control as measured by the Asthma Therapy Assessment Questionnaire (ATAQ) | 12 months post-intervention
  The Asthma Therapy Assessment Questionnaire (cATAQ) is a parent-report questionnaire; the symptom control subscale assesses children's asthma control (e.g., "wheezing or difficulty breathing") and shows good reliability and validity.

SECONDARY OUTCOMES:
Pediatric Quality of Life as measured by the Pediatric Quality of Life Inventory (PedsQL) Parent Report | Baseline
  The PedsQL is a brief and standardized questionnaire that assesses parents' perceptions of health-related quality of life for children with chronic health conditions. Parents will complete the parent report of child. Generic Core Scales of the PedsQL measure quality of life in physical, social, emotional and school domains (e.g., "it is hard for me to do chores around the house"; "it is hard to keep up when I play with other kids"), while the Asthma Module includes asthma-specific concerns related to symptoms and treatment (e.g., "I have trouble using my inhaler").
Pediatric Quality of Life as measured by the Pediatric Quality of Life Inventory (PedsQL) Parent Report | 1 week post-intervention
  The PedsQL is a brief and standardized questionnaire that assesses parents' perceptions of health-related quality of life for children with chronic health conditions. Parents will complete the parent report of child. Generic Core Scales of the PedsQL measure quality of life in physical, social, emotional and school domains (e.g., "it is hard for me to do chores around the house"; "it is hard to keep up when I play with other kids"), while the Asthma Module includes asthma-specific concerns related to symptoms and treatment (e.g., "I have trouble using my inhaler").
Pediatric Quality of Life as measured by the Pediatric Quality of Life Inventory (PedsQL) Parent Report | 6 months post-intervention
  The PedsQL is a brief and standardized questionnaire that assesses parents' perceptions of health-related quality of life for children with chronic health conditions. Parents will complete the parent report of child. Generic Core Scales of the PedsQL measure quality of life in physical, social, emotional and school domains (e.g., "it is hard for me to do chores around the house"; "it is hard to keep up when I play with other kids"), while the Asthma Module includes asthma-specific concerns related to symptoms and treatment (e.g., "I have trouble using my inhaler").
Pediatric Quality of Life as measured by the Pediatric Quality of Life Inventory (PedsQL) Parent Report | 12 months post-intervention
  The PedsQL is a brief and standardized questionnaire that assesses parents' perceptions of health-related quality of life for children with chronic health conditions. Parents will complete the parent report of child. Generic Core Scales of the PedsQL measure quality of life in physical, social, emotional and school domains (e.g., "it is hard for me to do chores around the house"; "it is hard to keep up when I play with other kids"), while the Asthma Module includes asthma-specific concerns related to symptoms and treatment (e.g., "I have trouble using my inhaler").
Pediatric Quality of Life as measured by the Pediatric Quality of Life Inventory (PedsQL) Child Self Report | Baseline
  The PedsQL is a brief and standardized questionnaire that assesses children's' perceptions of health-related quality of life for children with chronic health conditions. Children will complete the self-report version. Generic Core Scales of the PedsQL measure quality of life in physical, social, emotional and school domains (e.g., "it is hard for me to do chores around the house"; "it is hard to keep up when I play with other kids"), while the Asthma Module includes asthma-specific concerns related to symptoms and treatment (e.g., "I have trouble using my inhaler").
Pediatric Quality of Life as measured by the Pediatric Quality of Life Inventory (PedsQL) Child Self Report | 1 week post-intervention
  The PedsQL is a brief and standardized questionnaire that assesses children's' perceptions of health-related quality of life for children with chronic health conditions. Children will complete the self-report version. Generic Core Scales of the PedsQL measure quality of life in physical, social, emotional and school domains (e.g., "it is hard for me to do chores around the house"; "it is hard to keep up when I play with other kids"), while the Asthma Module includes asthma-specific concerns related to symptoms and treatment (e.g., "I have trouble using my inhaler").
Pediatric Quality of Life as measured by the Pediatric Quality of Life Inventory (PedsQL) Child Self Report | 6 months post-intervention
  The PedsQL is a brief and standardized questionnaire that assesses children's' perceptions of health-related quality of life for children with chronic health conditions. Children will complete the self-report version. Generic Core Scales of the PedsQL measure quality of life in physical, social, emotional and school domains (e.g., "it is hard for me to do chores around the house"; "it is hard to keep up when I play with other kids"), while the Asthma Module includes asthma-specific concerns related to symptoms and treatment (e.g., "I have trouble using my inhaler").
Pediatric Quality of Life as measured by the Pediatric Quality of Life Inventory (PedsQL) Child Self Report | 12 months post-intervention
  The PedsQL is a brief and standardized questionnaire that assesses children's' perceptions of health-related quality of life for children with chronic health conditions. Children will complete the self-report version. Generic Core Scales of the PedsQL measure quality of life in physical, social, emotional and school domains (e.g., "it is hard for me to do chores around the house"; "it is hard to keep up when I play with other kids"), while the Asthma Module includes asthma-specific concerns related to symptoms and treatment (e.g., "I have trouble using my inhaler").
Forced expiratory volume (FEV1) as measured by spirometry | Baseline
  FEV1 is the amount of air an individual can force from their lungs in one second and is a measure of lung function in pediatric asthma. FEV1 will be measured using a spirometer. Child participants will forcefully exhale their maximal amount of air in one second. Participants will perform 3-8 forced expiration maneuvers and the mean of the best three measurements will be used.
Forced expiratory volume (FEV1) as measured by spirometry | 1 week post-intervention
  FEV1 is the amount of air an individual can force from their lungs in one second and is a measure of lung function in pediatric asthma. FEV1 will be measured using a spirometer. Child participants will forcefully exhale their maximal amount of air in one second. Participants will perform 3-8 forced expiration maneuvers and the mean of the best three measurements will be used.
Forced expiratory volume (FEV1) as measured by spirometry | 6 months post-intervention
  FEV1 is the amount of air an individual can force from their lungs in one second and is a measure of lung function in pediatric asthma. FEV1 will be measured using a spirometer. Child participants will forcefully exhale their maximal amount of air in one second. Participants will perform 3-8 forced expiration maneuvers and the mean of the best three measurements will be used.
Forced expiratory volume (FEV1) as measured by spirometry | 12 months post-intervention
  FEV1 is the amount of air an individual can force from their lungs in one second and is a measure of lung function in pediatric asthma. FEV1 will be measured using a spirometer. Child participants will forcefully exhale their maximal amount of air in one second. Participants will perform 3-8 forced expiration maneuvers and the mean of the best three measurements will be used.
School attendance as measured by the Asthma Outcomes Questionnaire (AOQ) | Baseline
  Parent participants will complete an Asthma Outcomes Questionnaire (AOQ) designed for this study to assess their child's school absences related to asthma. Parent participants will report on the number of school absences in the past 6 months due to asthma.
School attendance as measured by the Asthma Outcomes Questionnaire (AOQ) | 1 week post-intervention
  Parent participants will complete an Asthma Outcomes Questionnaire (AOQ) designed for this study to assess their child's school absences related to asthma. Parent participants will report on the number of school absences in the past 6 months due to asthma.
School attendance as measured by the Asthma Outcomes Questionnaire (AOQ) | 6 months post-intervention
  Parent participants will complete an Asthma Outcomes Questionnaire (AOQ) designed for this study to assess their child's school absences related to asthma. Parent participants will report on the number of school absences in the past 6 months due to asthma.
School attendance as measured by the Asthma Outcomes Questionnaire (AOQ) | 12 months post-intervention
  Parent participants will complete an Asthma Outcomes Questionnaire (AOQ) designed for this study to assess their child's school absences related to asthma. Parent participants will report on the number of school absences in the past 6 months due to asthma.
Emergency Department visits as measured by the Asthma Outcomes Questionnaire (AOQ) | Baseline
  Parent participants will complete an Asthma Outcomes Questionnaire (AOQ) designed for this study to assess their child's emergency department visits related to asthma. Parent participants will report on the number of emergency department visits due to asthma in the past 6 months.
Emergency Department visits as measured by the Asthma Outcomes Questionnaire (AOQ) | 1 week post-intervention
  Parent participants will complete an Asthma Outcomes Questionnaire (AOQ) designed for this study to assess their child's emergency department visits related to asthma. Parent participants will report on the number of emergency department visits due to asthma in the past 6 months.
Emergency Department visits as measured by the Asthma Outcomes Questionnaire (AOQ) | 6 months post-intervention
  Parent participants will complete an Asthma Outcomes Questionnaire (AOQ) designed for this study to assess their child's emergency department visits related to asthma. Parent participants will report on the number of emergency department visits due to asthma in the past 6 months.
Emergency Department visits as measured by the Asthma Outcomes Questionnaire (AOQ) | 12 months post-intervention
  Parent participants will complete an Asthma Outcomes Questionnaire (AOQ) designed for this study to assess their child's emergency department visits related to asthma. Parent participants will report on the number of emergency department visits due to asthma in the past 6 months.
Hospitalizations as measured by the Asthma Outcomes Questionnaire (AOQ) | Baseline
  Parent participants will complete an Asthma Outcomes Questionnaire (AOQ) designed for this study to assess their child's hospitalizations related to asthma. Parent participants will report on the number of hospitalizations due to asthma in the past 6 months.
Hospitalizations as measured by the Asthma Outcomes Questionnaire (AOQ) | 1 week post-intervention
  Parent participants will complete an Asthma Outcomes Questionnaire (AOQ) designed for this study to assess their child's hospitalizations related to asthma. Parent participants will report on the number of hospitalizations due to asthma in the past 6 months.
Hospitalizations as measured by the Asthma Outcomes Questionnaire (AOQ) | 6 months post-intervention
  Parent participants will complete an Asthma Outcomes Questionnaire (AOQ) designed for this study to assess their child's hospitalizations related to asthma. Parent participants will report on the number of hospitalizations due to asthma in the past 6 months.
Hospitalizations as measured by the Asthma Outcomes Questionnaire (AOQ) | 12 months post-intervention
  Parent participants will complete an Asthma Outcomes Questionnaire (AOQ) designed for this study to assess their child's hospitalizations related to asthma. Parent participants will report on the number of hospitalizations due to asthma in the past 6 months.
Parent coping as measured by the Response to Stress Questionnaire (RSQ) | Baseline
  The Response to Stress Questionnaire - Pediatric Asthma Version (RSQ) is a questionnaire with parallel forms for youth self-report, parent report of child, and parent self-report, and yields scores for Primary Control Coping and Secondary Control Coping. The RSQ is appropriate for ages 9 and older, has been validated cross-culturally, has strong psychometric properties, and shows sensitivity to change as a mediator of coping skills interventions. Parents will complete the parent self-report form to assess their own coping.
Parent coping as measured by the Response to Stress Questionnaire (RSQ) | 1 week post-intervention
  The Response to Stress Questionnaire - Pediatric Asthma Version (RSQ) is a questionnaire with parallel forms for youth self-report, parent report of child, and parent self-report, and yields scores for Primary Control Coping and Secondary Control Coping. The RSQ is appropriate for ages 9 and older, has been validated cross-culturally, has strong psychometric properties, and shows sensitivity to change as a mediator of coping skills interventions. Parents will complete the parent self-report form to assess their own coping.
Parent coping as measured by the Response to Stress Questionnaire (RSQ) | 6 months post-intervention
  The Response to Stress Questionnaire - Pediatric Asthma Version (RSQ) is a questionnaire with parallel forms for youth self-report, parent report of child, and parent self-report, and yields scores for Primary Control Coping and Secondary Control Coping. The RSQ is appropriate for ages 9 and older, has been validated cross-culturally, has strong psychometric properties, and shows sensitivity to change as a mediator of coping skills interventions. Parents will complete the parent self-report form to assess their own coping.
Parent coping as measured by the Response to Stress Questionnaire (RSQ) | 12 months post-intervention
  The Response to Stress Questionnaire - Pediatric Asthma Version (RSQ) is a questionnaire with parallel forms for youth self-report, parent report of child, and parent self-report, and yields scores for Primary Control Coping and Secondary Control Coping. The RSQ is appropriate for ages 9 and older, has been validated cross-culturally, has strong psychometric properties, and shows sensitivity to change as a mediator of coping skills interventions. Parents will complete the parent self-report form to assess their own coping.
Parent report of child coping as measured by the Response to Stress Questionnaire (RSQ) | Baseline
  The Response to Stress Questionnaire - Pediatric Asthma Version (RSQ) is a questionnaire with parallel forms for youth self-report, parent report of child, and parent self-report, and yields scores for Primary Control Coping and Secondary Control Coping. The RSQ is appropriate for ages 9 and older, has been validated cross-culturally, has strong psychometric properties, and shows sensitivity to change as a mediator of coping skills interventions. Parents will complete the parent report of child form to assess their child's coping.
Parent report of child coping as measured by the Response to Stress Questionnaire (RSQ) | 1 week post-intervention
  The Response to Stress Questionnaire - Pediatric Asthma Version (RSQ) is a questionnaire with parallel forms for youth self-report, parent report of child, and parent self-report, and yields scores for Primary Control Coping and Secondary Control Coping. The RSQ is appropriate for ages 9 and older, has been validated cross-culturally, has strong psychometric properties, and shows sensitivity to change as a mediator of coping skills interventions. Parents will complete the parent report of child form to assess their child's coping.
Parent report of child coping as measured by the Response to Stress Questionnaire (RSQ) | 6 months post-intervention
  The Response to Stress Questionnaire - Pediatric Asthma Version (RSQ) is a questionnaire with parallel forms for youth self-report, parent report of child, and parent self-report, and yields scores for Primary Control Coping and Secondary Control Coping. The RSQ is appropriate for ages 9 and older, has been validated cross-culturally, has strong psychometric properties, and shows sensitivity to change as a mediator of coping skills interventions. Parents will complete the parent report of child form to assess their child's coping.
Parent report of child coping as measured by the Response to Stress Questionnaire (RSQ) | 12 months post-intervention
  The Response to Stress Questionnaire - Pediatric Asthma Version (RSQ) is a questionnaire with parallel forms for youth self-report, parent report of child, and parent self-report, and yields scores for Primary Control Coping and Secondary Control Coping. The RSQ is appropriate for ages 9 and older, has been validated cross-culturally, has strong psychometric properties, and shows sensitivity to change as a mediator of coping skills interventions. Parents will complete the parent report of child form to assess their child's coping.
Child self report of coping - Response to Stress Questionnaire (RSQ) | Baseline
  The Response to Stress Questionnaire - Pediatric Asthma Version (RSQ) is a questionnaire with parallel forms for youth self-report, parent report of child, and parent self-report, and yields scores for Primary Control Coping and Secondary Control Coping. The RSQ is appropriate for ages 9 and older, has been validated cross-culturally, has strong psychometric properties, and shows sensitivity to change as a mediator of coping skills interventions. Children will complete the child self-report form to assess their own coping.
Child self report of coping as measured by the Response to Stress Questionnaire (RSQ) | 1 week post-intervention
  The Response to Stress Questionnaire - Pediatric Asthma Version (RSQ) is a questionnaire with parallel forms for youth self-report, parent report of child, and parent self-report, and yields scores for Primary Control Coping and Secondary Control Coping. The RSQ is appropriate for ages 9 and older, has been validated cross-culturally, has strong psychometric properties, and shows sensitivity to change as a mediator of coping skills interventions. Children will complete the child self-report form to assess their own coping.
Child self report of coping as measured by the Response to Stress Questionnaire (RSQ) | 6 months post-intervention
  The Response to Stress Questionnaire - Pediatric Asthma Version (RSQ) is a questionnaire with parallel forms for youth self-report, parent report of child, and parent self-report, and yields scores for Primary Control Coping and Secondary Control Coping. The RSQ is appropriate for ages 9 and older, has been validated cross-culturally, has strong psychometric properties, and shows sensitivity to change as a mediator of coping skills interventions. Children will complete the child self-report form to assess their own coping.
Child self report of coping as measured by the Response to Stress Questionnaire (RSQ) | 12 months post-intervention
  The Response to Stress Questionnaire - Pediatric Asthma Version (RSQ) is a questionnaire with parallel forms for youth self-report, parent report of child, and parent self-report, and yields scores for Primary Control Coping and Secondary Control Coping. The RSQ is appropriate for ages 9 and older, has been validated cross-culturally, has strong psychometric properties, and shows sensitivity to change as a mediator of coping skills interventions. Children will complete the child self-report form to assess their own coping.
Family Asthma Management as measured by the Family Asthma Management Symptom Scale (FAMSS) | Baseline
  The Family Asthma Management Symptom Scale (FAMSS) is a semi-structured clinical interview administered jointly to youth (school-aged and older) and parents to assess family asthma management. The FAMSS captures adherence to asthma self-management behaviors such as symptom monitoring, trigger avoidance, and medication and healthcare use within the context of the family. It shows good reliability and is correlated with objective measures of management such as electronically monitored adherence.
Family Asthma Management as measured by the Family Asthma Management Symptom Scale (FAMSS) | 1 week post-intervention
  The Family Asthma Management Symptom Scale (FAMSS) is a semi-structured clinical interview administered jointly to youth (school-aged and older) and parents to assess family asthma management. The FAMSS captures adherence to asthma self-management behaviors such as symptom monitoring, trigger avoidance, and medication and healthcare use within the context of the family. It shows good reliability and is correlated with objective measures of management such as electronically monitored adherence.
Family Asthma Management as measured by the Family Asthma Management Symptom Scale (FAMSS) | 6 months post-intervention
  The Family Asthma Management Symptom Scale (FAMSS) is a semi-structured clinical interview administered jointly to youth (school-aged and older) and parents to assess family asthma management. The FAMSS captures adherence to asthma self-management behaviors such as symptom monitoring, trigger avoidance, and medication and healthcare use within the context of the family. It shows good reliability and is correlated with objective measures of management such as electronically monitored adherence.
Family Asthma Management as measured by the Family Asthma Management Symptom Scale (FAMSS) | 12 months post-intervention
  The Family Asthma Management Symptom Scale (FAMSS) is a semi-structured clinical interview administered jointly to youth (school-aged and older) and parents to assess family asthma management. The FAMSS captures adherence to asthma self-management behaviors such as symptom monitoring, trigger avoidance, and medication and healthcare use within the context of the family. It shows good reliability and is correlated with objective measures of management such as electronically monitored adherence.

CONTACTS AND LOCATIONS:
Overall Officials: Erin M Rodriguez, PhD, Principal Investigator — University of Texas at Austin
Locations (1):
- University of Texas at Austin, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rodriguez EM, Westcott S, Calderon MPY, Horner SD, Matsui EC, Dillard J, Fareed H, Camacho J. Study protocol for a randomized controlled trial of Adapt 2 Asthma (A2A), a culturally relevant coping skills and asthma management intervention for Latinx Families. Trials. 2024 Oct 22;25(1):706. doi: 10.1186/s13063-024-08531-w. PMID 39438915